CLINICAL TRIAL: NCT04711252
Title: SERENA-4: A Randomised, Multicentre, Double-Blind, Phase III Study of AZD9833 (an Oral SERD) Plus Palbociclib Versus Anastrozole Plus Palbociclib for the Treatment of Patients With Estrogen Receptor-Positive, HER2-Negative Advanced Breast Cancer Who Have Not Received Any Systemic Treatment for Advanced Disease
Brief Title: A Comparative Study of AZD9833 Plus Palbociclib Versus Anastrozole Plus Palbociclib in Patients With ER-Positive HER2 Negative Breast Cancer Who Have Not Received Any Systemic Treatment for Advanced Disease
Acronym: SERENA-4
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D8532C00001; 2020-002276-12 (EudraCT Number)
Record Dates: First submitted 2020-12-23; First posted 2021-01-15 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: ER-Positive HER2-Negative Breast Cancer
Keywords: Metastatic; Breast Neoplasms; Neoplasms by Site; Neoplasms; Breast Diseases; Skin Diseases; Hormones, Hormone Substitutes, and Hormone; Physiological Effects of Drugs; Randomised; Multicentre; Double-Blind; Phase III; AZD9833; Next Generation Oral SERD; Anastrozole; Palbociclib; Antagonists; Antineoplastic Agents; Estrogen Receptor Antagonists; Hormone Antagonists; camizestrant
MeSH Terms: conditions — Neoplasm Metastasis; Breast Neoplasms; Neoplasms by Site; Neoplasms; Breast Diseases; Skin Diseases | interventions — AZD9833; Anastrozole; palbociclib; Gonadotropin-Releasing Hormone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AZD9833 + palbociclib (Experimental): The patients will receive AZD9833 (75 mg, PO, once daily) + palbociclib (PO, once daily, 125 mg for 21 consecutive days followed by 7 days off treatment) + anastrozole placebo (1 mg, PO, once daily)
  Interventions: Drug: AZD9833; Drug: Anastrozole placebo; Drug: Palbociclib; Drug: Luteinizing hormone-releasing hormone (LHRH) agonist
- Anastrozole + palbociclib (Active Comparator): The patients will recieve Anastrozole (1 mg, PO, once daily) + palbociclib (PO, once daily, 125 mg for 21 consecutive days followed by 7 days off treatment) + AZD9833 placebo (PO, once daily)
  Interventions: Drug: Anastrozole; Drug: AZD9833 placebo; Drug: Palbociclib; Drug: Luteinizing hormone-releasing hormone (LHRH) agonist

INTERVENTIONS:
Drug: AZD9833 — Dosage formulation: AZD9833 tablets will be administered orally
  Arms: AZD9833 + palbociclib
Drug: Anastrozole — Dosage formulation: Anastrozole tablets will be administered orally.
  Arms: Anastrozole + palbociclib
Drug: Anastrozole placebo — Dosage formulation: anastrozole placebo tablets will be administrated orally.
  Arms: AZD9833 + palbociclib
Drug: AZD9833 placebo — Dosage formulation: AZD9833 placebo tablets will be administrated orally.
  Arms: Anastrozole + palbociclib
Drug: Palbociclib — Dosage formulation: palbociclib tablets/capsules will be administered orally
Drug: Luteinizing hormone-releasing hormone (LHRH) agonist — Men (when medically applicable) and pre- or peri-menopausal women are required to receive a monthly LHRH agonist.

SUMMARY:
The study is intended to show superiority of AZD9833 in combination with palbociclib (a CDK4/6 inhibitor) versus anastrozole (an aromatase inhibitor) and palbociclib as the initial treatment of patients with hormone receptor-positive (ER-positive), human epidermal growth factor 2-negative (HER2-negative) advanced/metastatic breast cancer.

INFORMATION FOR TRIAL PARTICIPANTS

In this trial, the researchers will look at how well camizestrant with palbociclib works, compared with anastrozole with palbociclib, in participants with breast cancer that has either spread into other parts of the body at the time of diagnosis, or has come back after at least 2 years of standard endocrine treatment.

Participants in this trial will have breast cancer that has ER proteins but does not have overexpression of HER2 protein.

DETAILED DESCRIPTION:
A Randomised, Multicentre, Double-Blind, Phase III study will evaluate the safety and efficacy of AZD9833 (next generation oral SERD) in combination with palbociclib versus anastrozole in combination with palbociclib for the treatment of patients with ER-positive breast cancer. The goal of the study is to demonstrate superiority of AZD9833 over anastrozole in the context of combination with palbociclib in first line setting.

INFORMATION FOR TRIAL PARTICIPANTS

Researchers are looking for a better way to treat breast cancer.

In people with cancer, some cells have grown out of control to form tumours.

The trial drugs palbociclib, camizestrant, and anastrozole are designed to work by blocking the cancer's ability to grow. Camizestrant is also called AZD9833. Palbociclib and anastrozole are already available as treatments for people with certain type of breast cancer.

In this trial, the researchers want to find out how well taking camizestrant with palbociclib, or anastrozole with palbociclib, works in participants with breast cancer that has ER proteins but does not have overexpression of HER2 protein.

The researchers will look at which trial treatments help the participants live longer with cancer before it gets worse.

The trial will split participants into 2 groups:

* Participants in Group 1 will take camizestrant, palbociclib, and a placebo matched with anastrazole.
* Participants in Group 2 will take anastrozole, palbociclib, , and a placebo matched with camizestrant.

A placebo looks like a treatment but does not have any medicine in it.

A computer program will be used to randomly choose the treatments each participant gets. This helps make sure the groups are chosen fairly. Researchers do this so that comparing the results of each treatment will be as accurate as possible.

The participants will take their trial treatments in periods called "cycles". Each cycle will last 28 days. During each cycle, the participants will take:

* camizestrant or anastrozole once daily by mouth
* palbociclib once daily by mouth for 21 days. Then, they will not take any palbociclib for 7 days

Some participants will also get either goserelin or leuprorelin once every month. Participants could get goserelin or leuprorelin if:

* They are medically determined yet to reach menopause status
* They are male

They will get this treatment as an injection under the skin or into a muscle. Goserelin and leuprorelin work by decreasing the amount of sex hormones made by the body which will lead to reduction of ER production. This can help stop breast cancer from growing.

Participants will take trial treatment until the cancer gets worse or they leave the trial.

Participants will visit their trial site several times throughout the trial. At these visits, the trial doctors will check the health of the participants. They will also take blood samples and do scans of the participants' tumors.

ELIGIBILITY:
INCLUSION CRITERIA

Full list of inclusion criteria

* Pre-/peri-menopausal women or men can be enrolled if amenable to be treated with concomitant, approved LHRH agonists for the duration of the study treatment.
* De novo Stage 4 disease, or recurrence from early stage disease after at least 24 months of standard adjuvant endocrine therapy. Note that at least 12 months must have elapsed since the patient's last dose of adjuvant AI therapy without disease progression on treatment. Note that a 2-week washout period is required after the last dose of tamoxifen prior to randomisation.
* Histologically or cytologically documented diagnosis of ER+, HER2-negative breast cancer based on local laboratory results.
* Previously untreated with any systemic anti-cancer therapy for their locoregionally recurrent or metastatic ER+ disease.
* Measurable disease as defined per RECIST v.1.1 OR at least one lytic or mixed (lytic + sclerotic) bone lesion with a soft tissue component that can be assessed by CT or MRI.
* Eastern Cooperative Oncology Group performance status of 0 or 1.
* Adequate organ and marrow function.
* Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

INFORMATION FOR TRIAL PARTICIPANTS

Participants can join the trial if they:

* Have breast cancer that cannot be treated with surgery or radiation
* Have breast cancer that has already spread into other parts of the body at the time of diagnosis, or has come back after at least 2 years of a standard endocrine treatment
* Have ER proteins but not overexpression of HER2 protein in their tumors
* Have never received any type of cancer therapy that affects the whole body for advanced breast cancer
* Are able to do their daily activities

EXCLUSION CRITERIA

Full list of exclusion criteria

* Previous neoadjuvant or adjuvant treatment with an AI treatment +/- CDK4/6 inhibitor with disease recurrence while on or within 12 months of completing treatment.
* Prior exposure to AZD9833, other investigational SERDs/endocrine agents or fulvestrant.
* Participation in another clinical study with a study treatment or investigational medicinal device administered in the last 4 weeks prior to randomization or concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study.
* Advanced, symptomatic, visceral spread, that are at risk of life-threatening complications in the short term and/or impending visceral crisis
* Known active uncontrolled or symptomatic CNS metastases, carcinomatous meningitis, or leptomeningeal disease.
* Any clinically important and symptomatic heart disease .
* Currently pregnant (confirmed with positive pregnancy test) or breast-feeding.
* As judged by the investigator, any evidence of diseases (such as severe or uncontrolled systemic diseases, renal transplant and active bleeding diseases) which, in the investigator's opinion, makes it undesirable for the participant to participate in the study or that would jeopardize compliance with the protocol.
* Any concurrent anti-cancer treatment.
* Active infection including tuberculosis, HBV and HCV.

INFORMATION FOR TRIAL PARTICIPANTS

Participants cannot join the trial if they:

* Have uncontrolled cancer that has spread to the brain or the spinal cord
* Have received certain treatments for cancer in the past but the cancer came back within 1 year
* Had certain types of tumors in the past, which the study doctors think could come back
* Are currently taking any treatment for cancer or are taking medications or supplements that affect certain proteins in the body
* Have any major health problem, infection, or surgery that could make it difficult or dangerous to participate in this trial, such as tuberculosis, HIV, heart problems, or a kidney transplant

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1370 (Actual)
Dates: Start 2021-01-28 (Actual); Primary Completion 2026-08-24 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) assessed by the Investigator as defined by response evaluation criteria in solid tumors (RECIST) version 1.1 | From randomization until progression per RECIST 1.1 as assessed by the investigator at local site or death due to any cause (up to 5 years)
  PFS is defined as the time from randomization to objective disease progression (as assessed by RECIST) or death.

SECONDARY OUTCOMES:
Overall survival (OS) | From randomization until the date of death due to any cause (up to 8 years)
  The OS is defined as the time from randomization to death due to any cause.
Second progression-free survival (PFS2) | From randomization to the earliest of the progression event (following the initial progression), subsequent to first subsequent therapy or death (up to 5 years)
  Time to second progression or death (PFS2) will be defined as the time from randomisation to the earliest of the progression event (following the initial progression), subsequent to first subsequent therapy or death.
Objective response rate (ORR) assessed by the Investigator as defined by RECIST version 1.1 | From randomization until a response or in the absence of a response from randomization up until progression, or the last evaluable assessment in the absence of progression (up to 5 years)
  ORR is defined as the proportion of patients who have a CR or partial response, as determined by the investigator at local site per RECIST 1.1.
Duration of response (DoR) assessed by the Investigator as defined by RECIST version 1.1 | From the date of first documented response until date of documented progression per RECIST 1.1 as assessed by the investigator at local site or death due to any cause (up to 5 years)
  The DoR will be defined as the time from the date of first documented response until date of documented progression or death in the absence of disease progression.
Time to chemotherapy (TTC) | From randomization until the earlier of the start date of chemotherapy or death due to any cause (up to 5 years)
  Time to chemotherapy is defined as the time from randomization until the earlier of the start date of chemotherapy or death due to any cause.
Time to first subsequent anti-cancer therapy (TFST) | From randomization until the earlier of start date of the first subsequent anti-cancer therapy after discontinuation of randomized treatment, or death due to any cause (up to 5 years)
  TFST is defined as time from randomization until the earlier of start date of the first subsequent anti-cancer therapy after discontinuation of randomized treatment, or death due to any cause.
Clinical benefit rate at 24 weeks (CBR24) | At least 23 weeks after randomisation
  CBR at 24 weeks is defined as the percentage of participants who have a complete response (CR) or partial response or who have stable disease (SD) per RECIST 1.1 as assessed by the investigator at local site for at least 23 weeks after randomization (to allow for an early assessment within the assessment window).
Time to second subsequent therapy (TSST) | From randomization until the earlier of start date of the second subsequent anti-cancer therapy after discontinuation of first subsequent treatment, or death due to any cause (up to 5 years)
  TSST is defined as time from randomization until the earlier of start date of the second subsequent anti-cancer therapy after discontinuation of first subsequent treatment, or death due to any cause.
Plasma concentration of AZD9833 at specified timepoints | on Day 15
  To assess the steady state PK of AZD9833 in combination with palbociclib in all participants who receive at least one dose of AZD9833 per the protocol, for whom there are at least one reportable PK concentration.
Change from baseline in EORTC QLQ-C30 scale scores | From baseline to 24 weeks post progression (up to approximately 5 years)
  Change from baseline in EORTC QLQ-C30 scale scores for each patient at each post-baseline visit. The comparison will include all randomised patients, as randomised, with baseline and at least one post-baseline visit score for the scale score.
Change from baseline in EORTC QLQ-BR45 scale scores | From baseline to 24 weeks post progression (up to approximately 5 years)
  Change from baseline in EORTC QLQ-BR45 scale scores for each patient at each post-baseline visit. The comparison will include all randomised patients, as randomised, with baseline and at least one post-baseline visit score for the scale score.

CONTACTS AND LOCATIONS:
Locations (216):
- United States (28):
  - Research Site, Mobile, Alabama
  - Research Site, Springdale, Arkansas
  - Research Site, Harbor City, California
  - Research Site, Solvang, California
  - Research Site, Lone Tree, Colorado
  - Research Site, Fort Myers, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Indianapolis, Indiana
  - Research Site, Baton Rouge, Louisiana
  - Research Site, Silver Spring, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Hattiesburg, Mississippi
  - Research Site, Omaha, Nebraska
  - Research Site, Cincinnati, Ohio
  - Research Site, Portland, Oregon
  - Research Site, West Columbia, South Carolina
  - Research Site, Sioux Falls, South Dakota
  - Research Site, Chattanooga, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Houston, Texas
  - Research Site, Tyler, Texas
  - Research Site, Fairfax, Virginia
  - Research Site, Kennewick, Washington
  - Research Site, Renton, Washington
  - Research Site, Morgantown, West Virginia
- Austria (3):
  - Research Site, Feldkirch
  - Research Site, Salzburg
  - Research Site, Vienna
- Belgium (7):
  - Research Site, Anderlecht
  - Research Site, Edegem
  - Research Site, Ghent
  - Research Site, Leuven
  - Research Site, Liège
  - Research Site, Namur
  - Research Site, Sint-Niklaas
- Bulgaria (3):
  - Research Site, Plovdiv
  - Research Site, Shumen
  - Research Site, Sofia
- Canada (6):
  - Research Site, Edmonton, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Kitchener, Ontario
  - Research Site, London, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal
- Chile (3):
  - Research Site, Concepción
  - Research Site, La Serena
  - Research Site, Santiago
- China (24):
  - Research Site, Baoding
  - Research Site, Beijing
  - Research Site, Bengbu
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Dalian
  - Research Site, Guangzhou
  - Research Site, Guiyang
  - Research Site, Haikou
  - Research Site, Hangzhou
  - Research Site, Hefei
  - Research Site, Jinan
  - Research Site, Lanzhou
  - Research Site, Linyi
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Tianjin
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Zhengzhou
- Czechia (4):
  - Research Site, Hořovice
  - Research Site, Hradec Králové
  - Research Site, Nový Jičín
  - Research Site, Prague
- France (13):
  - Research Site, Besançon
  - Research Site, Bordeaux
  - Research Site, Brest
  - Research Site, Caen
  - Research Site, Dijon
  - Research Site, Le Mans
  - Research Site, Lille
  - Research Site, Montpellier
  - Research Site, Pierre-Bénite
  - Research Site, Plerin SUR MER
  - Research Site, Saint-Cloud
  - Research Site, Vandœuvre-lès-Nancy
  - Research Site, Villejuif
- Germany (9):
  - Research Site, Berlin
  - Research Site, Dessau-RoBlau
  - Research Site, Essen
  - Research Site, Freiburg im Breisgau
  - Research Site, Mönchengladbach
  - Research Site, München
  - Research Site, Münster
  - Research Site, Regensburg
  - Research Site, Velbert
- Hungary (6):
  - Research Site, Budapest
  - Research Site, Győr
  - Research Site, Miskolc
  - Research Site, Nyíregyháza
  - Research Site, Szekszárd
  - Research Site, Zalaegerszeg
- India (11):
  - Research Site, Ahmedabad
  - Research Site, Calicut
  - Research Site, Delhi
  - Research Site, Faridabad
  - Research Site, Gūrgaon
  - Research Site, Karamsad
  - Research Site, Kolkata
  - Research Site, Madurai
  - Research Site, Nagpur
  - Research Site, Nashik
  - Research Site, New Delhi
- Italy (11):
  - Research Site, Bergamo
  - Research Site, Florence
  - Research Site, Milan
  - Research Site, Modena
  - Research Site, Napoli
  - Research Site, Novara
  - Research Site, Padua
  - Research Site, Parma
  - Research Site, Prato
  - Research Site, Roma
  - Research Site, Rozzano
- Japan (25):
  - Research Site, Chiba
  - Research Site, Chūōku
  - Research Site, Hidaka-shi
  - Research Site, Hirakata-shi
  - Research Site, Isehara-shi
  - Research Site, Kitaadachi-gun
  - Research Site, Kōtoku
  - Research Site, Kumamoto
  - Research Site, Kurashiki Shi
  - Research Site, Kurume-shi
  - Research Site, Kyoto
  - Research Site, Nagoya
  - Research Site, Nishinomiya-shi
  - Research Site, Osaka
  - Research Site, Ota-shi
  - Research Site, Sapporo
  - Research Site, Sendai
  - Research Site, Shimotsuke-shi
  - Research Site, Shinagawa-ku
  - Research Site, Shinjuku-ku
  - Research Site, Suita-shi
  - Research Site, Takasaki-shi
  - Research Site, Tsu
  - Research Site, Tsukuba
  - Research Site, Yokohama
- Malaysia (5):
  - Research Site, George Town
  - Research Site, Johor Bahru
  - Research Site, Kuala Lumpur
  - Research Site, Kuala Selangor
  - Research Site, Kuching
- Mexico (6):
  - Research Site, Del. Cuauhtemoc
  - Research Site, Estado de México
  - Research Site, La Paz
  - Research Site, Mexico City
  - Research Site, Monterrey
  - Research Site, Puebla City
- Norway (2):
  - Research Site, Drammen
  - Research Site, Oslo
- Poland (7):
  - Research Site, Gdynia
  - Research Site, Konin
  - Research Site, Koszalin
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Olsztyn
  - Research Site, Poznan
- Portugal (6):
  - Research Site, Braga
  - Research Site, Guimarães
  - Research Site, Lisbon
  - Research Site, Loures
  - Research Site, Porto
  - Research Site, Vila Nova de Gaia
- Russia (4):
  - Research Site, Kaluga
  - Research Site, Kislino Village, Ryshkovsky Ru
  - Research Site, Moscow
  - Research Site, Saint Petersburg
- Slovakia (4):
  - Research Site, Banská Bystrica
  - Research Site, Bratislava
  - Research Site, Prešov
  - Research Site, Trenčín
- South Korea (4):
  - Research Site, Busan
  - Research Site, Daegu
  - Research Site, Goyang-si
  - Research Site, Seoul
- Spain (9):
  - Research Site, Barcelona
  - Research Site, Jaén
  - Research Site, Lleida
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Pamplona
  - Research Site, Santander
  - Research Site, Seville
  - Research Site, Valencia
- Switzerland (2):
  - Research Site, Liestal
  - Research Site, Zurich
- Taiwan (5):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Turkey (Türkiye) (4):
  - Research Site, Adana
  - Research Site, Ankara
  - Research Site, Izmir
  - Research Site, Kayseri
- United Kingdom (5):
  - Research Site, Cambridge
  - Research Site, Colchester
  - Research Site, Leeds
  - Research Site, Nottingham
  - Research Site, Surrey

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: BreastCancerStudyLocator.com — https://breastcancerstudylocator.com/